CLINICAL TRIAL: NCT05912231
Title: Proton Versus Photon Ultrahypofractionated Radiation Therapy and Its Impact on Normal Tissue
Brief Title: Ultrahypofractionation and Normal Tissue Toxicity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Rachel Beth Jimenez, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-182; P01CA261669 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Cancer Stage II; Breast Cancer Stage III; Myocardial Fibrosis
Keywords: Radiation Therapy; Photon Radiation Therapy; XRT; Proton Beam Radiation Therapy; PBT; Breast Cancer; Breast Cancer Female; Breast Cancer Stage II; Breast Cancer Stage III; Myocardial Fibrosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Accelerated Proton Beam Radiation Therapy (PBT) Group (Experimental): Participants will be randomized 1:1 to XRT group and stratified by receipt of chemotherapy and cardiac risk factors and will complete:
  * Cardiac MRI and blood tests within 1 month prior to start of radiation therapy.
  * Radiation therapy 1x daily for 5 days over 1 week.
  * End of radiation therapy visit with blood tests.
  * 6 month follow up visit with cardiac MRI, blood tests, questionnaires, and photographic imaging.
  * 12 month follow up visit with questionnaires and photographic imaging.
  Interventions: Radiation: Accelerated Proton Beam Radiation Therapy (PBT)
- Accelerated Photon Radiation Therapy (XRT) Group (Experimental): Participants will be randomized 1:1 to XRT group and stratified by receipt of chemotherapy and cardiac risk factors and will complete:
  * Cardiac MRI and blood tests within 1 month prior to start of radiation therapy.
  * Radiation therapy 1x daily for 5 days over 1 week.
  * End of radiation therapy visit with blood tests.
  * 6 month follow up visit with cardiac MRI, blood tests, questionnaires, and photographic imaging.
  * 12 month follow up visit with questionnaires and photographic imaging.
  Interventions: Radiation: Accelerated Photon Radiation Therapy (XRT)

INTERVENTIONS:
Radiation: Accelerated Proton Beam Radiation Therapy (PBT) — per protocol
  Arms: Accelerated Proton Beam Radiation Therapy (PBT) Group
Radiation: Accelerated Photon Radiation Therapy (XRT) — per protocol
  Arms: Accelerated Photon Radiation Therapy (XRT) Group

SUMMARY:
This research is being done to see if proton beam radiation therapy (PBT) results in fewer changes to a participant's heart measured with MRI-imaging than conventional or "photon" radiation therapy (XRT) for participants with non-metastatic left sided breast cancer.

The names of the two study groups in this research study are:

* Proton Radiation Therapy (PBT)
* Conventional or "Photon" Radiation Therapy (XRT)

DETAILED DESCRIPTION:
This is a randomized phase II trial comparing participants with stage II-III breast cancer treated with accelerated Proton Beam Radiation Therapy (PBT) versus accelerated conventional photon radiation therapy (XRT) inclusive of the regional lymph nodes.

Participants will be randomized into one of two study groups: proton beam radiation therapy versus photon radiation therapy. Randomization means that participants are put into a group by chance.

Study procedures includes screening for eligibility, study treatment visits, Cardiac Magnetic Resonance Imaging (MRI), blood tests, and questionnaires.

The National Cancer Institute, American Society of Clinical Oncology, and Claflin Grant are supporting this research by providing funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Non-metastatic Breast Cancer patients who are scheduled to receive conventional left-sided or bilateral breast/chest wall RT inclusive of treatment to the internal mammary lymph nodes (IMNs)
* Prior chemotherapy is permitted
* Ability to understand and the willingness to sign a written informed consent document
* No contraindication to MRI
* Patients with right-sided breast cancer or patients with left-sided patients not requiring treatment to the IMNs, but where cardiac anatomy is determined to be unfavorable by the study PI, will be considered eligible.

Exclusion Criteria:

* Person who is pregnant or breastfeeding.
* Patients receiving any other investigational agent will not be excluded from study eligibility, unless the patient is already enrolled in an interventional study evaluating cardiac toxicity. No cytotoxic therapy or radiotherapy may be used during radiation therapy.
* Contra-indication to gadolinium contrast (e.g., chronic kidney disease)
* Contra-indication to radiotherapy (e.g., scleroderma, p53 mutation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All women of all races and ethnic groups are eligible for this trial.
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial Fibrosis from Baseline in Proton Beam Radiation Therapy (PBT) | Up to 7 months (pre-treatment period to 6 month follow up)
  The primary outcome is to determine whether participants who receive accelerated PBT show no increase in myocardial fibrosis on Cardiac MRI (CMR) compared to an estimated 4% increase in extracellular matrix volume fraction (ECV) in participants who receive accelerated XRT. CMR will be performed using a 3T system (Skyra, Siemens). The T1 phase on MRI will be used to measure ECV.

SECONDARY OUTCOMES:
Change in Global Longitudinal Strain (GLS) on CMR from Baseline | Up to 7 months (pre-treatment period to 6 month follow up)
  GLS will be measured using feature tracking from the Steady-state free precession (SSFP) MRI cine images (Medis Suite, Leiden).
Stability of Cardiac Biomarkers from Baseline | Up to 7 months (pre-treatment period to 6 month follow up)
  Cardiac Biomarkers will be measured using enzyme-linked immunoassay (ELISA).
Body Image Evaluation | Up to 13 months (pre-treatment period to 12 month follow up)
  Assessed by photographic imaging of the breast, chest wall and reconstructed breast, the Breast Q: Mastectomy Module (Postoperative) 2.0, the Breast Q: Reconstruction Module (Postoperative) 2.0, and the Breast-Q: Breast Conserving Therapy Module (Postoperative) 2.0 questionnaires which are rigorous patient-report outcome measures. Modules grade Quality of Life (QOL) and Satisfaction Domains related to post-operative care and experiences. All BREAST-Q scales are transformed into scores that range from 0-100. T. A higher score means greater satisfaction or better QOL (depending on the scale).
Change in Shoulder Function from Baseline | Up to 13 months (pre-treatment period to 12 month follow up)
  Assessed by the Thoracic Focused Assessment with Sonography for Trauma, Triage, and Tracking (TFAST), the Penn Shoulder Scale (PSS), and the Disabilities of the Arm, Shoulder and Hand (DASH) Shoulder Function Scale. TFAST is an objective and highly reproducible functional assessment tool of the arm and shoulder. The PSS is a patient-reported outcome tool which provides a shoulder-specific metric and distinguishes between finer levels of functioning. Scores range from 0 to 100 with a score of 100 indicating low pain, high satisfaction, and high function. DASH is a 30-item, validated, patient-reported scale that captures upper extremity functionality and mobility and maintains high construct validity and responsiveness in the breast cancer population. Questions are graded on a Likert scale with scores ranging from "1" Strongly Disagree to "5" Strongly Agree, where a cumulative score of 0 is graded no disability and 100 is most severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jimenez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation